CLINICAL TRIAL: NCT06945796
Title: ACT-ED: ACT-Based Eating Disorder Prevention Program
Brief Title: ACT-ED: Accessibility and Feasibility of an Acceptance and Commitment Therapy (ACT)-Based Eating Disorder Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Haldun University (Other)
Responsible Party: Principal Investigator, Emine Serra Nebati, Principal Investigator, Ibn Haldun University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024/09-08
Record Dates: First submitted 2025-04-11; First posted 2025-04-25 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: Eating Disorders Symptoms; Eating Pathology; Disordered Eating Behaviors
Keywords: disordered eating; eating pathology; prevention; eating disorders; early intervention
MeSH Terms: conditions — Disordered Eating Behavior; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group intervention (Experimental): ACT-based online group intervention. 4 sessions of 1.5 hours, held once a week
  Interventions: Other: ACT based eating disorder prevention program

INTERVENTIONS:
Other: ACT based eating disorder prevention program — This intervention protocol was developed specifically for women who have body dissatisfaction and disordered eating behaviors. Based on the psychological flexibility model (hexaflex), it is designed to improve people's body image flexibility using Acceptance and Commitment Therapy techniques.
  Interventions related to the dimensions of the hexaflex were made during each session. The first session covers values and goal setting. The second session includes creative hopelessness, acceptance, and self-compassion. The third session covers defusion and mindfulness. The last session focuses on self-as-context exercises and the combined use of skills for committed action.
  Other Names: ACT-ED

SUMMARY:
The goal of this clinical trial is to investigate the accessibility and feasibility of an online group prevention program developed for women at risk for eating disorders. Also, to conduct a preliminary analysis of treatment efficacy. The main questions it aims to answer are:

Does ACT-ED an acceptable intervention for women at risk for eating disorders? Does intervention result in reduced eating pathology?

Participants will:

Join the online, 4-session ACT-based group program Fill the measures at Pre-test, post-test and follow-up assessment

ELIGIBILITY:
Inclusion Criteria:

* Being a woman aged 18 years or older
* Exhibiting disordered eating behaviors (EDE-Q score ≥ 3.03)
* Experiencing body dissatisfaction (BSQ-34 score ≥ 110)

Exclusion Criteria:

* Current or past diagnosis/treatment for an eating disorder
* Currently receiving psychotherapy
* Currently receiving psychiatric medication (not excluded if there has been no change in treatment in the last 6 months)
* Having chronic psychiatric disorders (e.g. psychosis)
* Having a substance addiction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — biological females
Enrollment: 5 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Disordered eating, assessed by the Turkish form of the Eating disorder examination questionnaire (EDE-Q) | Baseline (pretest), week 4(posttest), 1-month follow-up
  Disordered eating is a risk factor for eating disorders. In a prevalence study conducted in Türkiye, individuals with EDE-Q scores of 3.03 and above were defined as a high-risk group (Deveci, 2020). In this study, EDE-Q scores were assessed for inclusion criteria during enrollment. Additionally, changes in EDE-Q scores are assessed at post-test and follow-up to assess treatment effect.

SECONDARY OUTCOMES:
Body dissatisfaction, assessed by the Turkish form of Body shape Questionnaire (BSQ) | Baseline (pretest), week 4(posttest), 1-month follow-up
  A total score of the questionnaire can be in the range of 34 to 204 where total score lower than 110 represents no concern, a total score between 110 and 137 represents mild concern, a total score between 138 and 166 represents moderate concern, and a total score higher than 167 represent severe concern. In this study, EDE-Q scores were assessed for inclusion criteria during enrollment; participants scores of 110 and above are included. Additionally, changes in EDE-Q scores are assessed at post-test and follow-up.
Body image flexibility, assessed by the Turkish form of the Body Image Acceptance and Action Questionnaire (BI-AAQ) | Baseline (pretest), week 4(posttest), 1-month follow-up
  Body image flexibility (BIF) is a construct derived from the psychological flexibility model. BIF is defined as the capacity to experience perceptions, sensations, feelings, thoughts, and beliefs related to one's body without avoidance while acting in alignment with personal values. The BI-AAQ consists of 12 items; higher scores indicate lower BIF and increased body image inflexibility. In this study, this scale would be used to assess how one's relation with body image-related internal experiences changes after the prevention program.
Psychological flexibility, assessed by Acceptance and Action Questionnaire (AAQ-II) | Baseline (pretest), week 4(posttest), 1-month follow-up
  The AAQ-II is designed to assess psychological flexibility defined as the capacity to be in contact with the present moment, fully aware of one's thoughts, emotions, and sensations. Higher scores indicate decreased psychological flexibility and increased experiential avoidance. In this study, the scale was used to assess changes in the general psychological flexibility.
Present moment awareness, assessed by the Turkish form of the Freiburg Mindfulness Inventory (FMI) | Baseline (pretest), week 4(posttest), 1-month follow-up
  Present moment awareness is one of the dimensions of the psychological flexibility model. It is defined as the ability to fully engage with the present moment. Higher scores indicate better present moment awareness. In future studies, it is desired to examine which dimension of the psychological flexibility model has an effect on the treatment outcome. In this study, FMI was used to test its suitability in measuring change in this intervention.
Contextual Self, assessed by the Turkish form of the Self-As-Context Scale (SACS) | Baseline (pretest), week 4(posttest), 1-month follow-up
  Contextual Self is one of the dimensions of the psychological flexibility model. It is defined as one's ability to view himself with a broader perspective. Higher scores indicate improved contextual self. In future studies, it is desired to examine which dimension of the psychological flexibility model has an effect on the treatment outcome. In this study, SACS was used to test its suitability in measuring change in this intervention.
Defusion, assessed by the Turkish form of the Cognitive Fusion Scale (CFS) | Baseline (pretest), week 4(posttest), 1-month follow-up
  Defusion is one of the dimensions of the psychological flexibility model. It is defined as one's ability to separate himself from his thoughts. Higher scores indicate fusion, which is the opposite of defusion. In future studies, it is desired to examine which dimension of the psychological flexibility model has an effect on the treatment outcome. In this study, SACS was used to test its suitability in measuring change in this intervention.
Personality beliefs, assessed by the Turkish form of the Personality Beliefs Questionnaire- Short Form (PBQ-SF) | Baseline (pretest), week 4(posttest), 1-month follow-up
  Obsessive-compulsive personality disorder and borderline personality disorder are the most common personality disorders in eating disorders. PBQ is designed to assess dysfunctional personality beliefs, and higher scores on a subscale indicate stronger dysfunctional beliefs related to the corresponding personality.
  In future studies, it is desired to examine how the personality beliefs are affected by the prevention program. In this study, PBQ-SF was used to test its suitability in measuring change in personality beliefs by this intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Serra Nebati, Principal Investigator — Ibn Haldun University
Locations (1):
- Ibn Haldun University Psychotherapy Application and Research Center (IPAM), Istanbul, Basaksehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to confidentiality concerns and ethical considerations.